CLINICAL TRIAL: NCT04801706
Title: Association of Ultrasonographic Parameters With FIGO Clinical Grading System for Placenta Accreta Spectrum: A Prospective Cohort Study
Brief Title: Association of Ultrasonographic Parameters With FIGO Clinical Grading System for Placenta Accreta Spectrum
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Sayed Reyad, Assiut University, Women Health Hospital, Assiut University
Other Study IDs: Prenatal US and clinical FIGO
Record Dates: First submitted 2021-03-10; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Placenta Accreta, Unspecified Trimester
MeSH Terms: conditions — Placenta Accreta | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound — Association of each ultrasonographic parameter with FIGO clinical grading of placenta accreta and with histopathological diagnosis of placenta accreta in hysterectomy specimens

SUMMARY:
To evaluate the association of ultrasonographic parameters suggestive of placenta accreta with intraoperative clinical diagnosis of placenta accreta according to the the clinical grading system for placenta accreta spectrum (PAS) disorders proposed recently by FIGO and histopathological diagnosis of placenta accreta in hysterectomy specimens

DETAILED DESCRIPTION:
Evaluation of the association of ultrasonographic parameters suggestive of placenta accreta with intraoperative clinical diagnosis of placenta accreta according to the the clinical grading system for placenta accreta spectrum (PAS) disorders proposed recently by FIGO and histopathological diagnosis of placenta accreta in hysterectomy specimens The following ultrasound items will be examined: number and viability of fetuses, amniotic fluid assessment, fetal biometries, fetal gender if possible, fetal presentation, Estimated fetal weight using Hadlock formula, Umbilical Artery Pulsatility Index (UA PI) measured from an automated/manual trace of at least three consecutive waveforms of the relevant vessel in the absence of fetal breathing movements or uterine contractions. The UA PI will be recorded from a free-floating section of cord.

Next step the investigators will look for suggestive ultrasound parameters of placenta accreta including:

1. Location of placenta: Placenta previa anterior / posterior / totally covering the internal cervical os.
2. Lacunae staging according to Finberg and Williams as follows: grade 0, none seen; grade 1, 1-3 present and generally small; grade 2, 4-6 present and tending to be larger and more irregular; grade 3, many throughout the placenta and appearing large and bizarre.
3. Loss of the clear zone, defined as loss or irregularity of the hypoechoic plane in the myometrium underneath the placental bed
4. Bladder wall interruption, defined as loss or interruption of the bright bladder wall (hyperechoic band or 'line' between the uterine serosa and bladder lumen)
5. Uterovescical hypervascularity, defined as a striking amount of color Doppler signal seen between the myometrium and the posterior wall of the bladder, including vessels appearing to extend from the placenta, across the myometrium and beyond the serosa, into the bladder or other organs, often running perpendicular to the myometrium.
6. Increased vascularity in the parametrial region, defined as the presence of hypervascularity extending beyond the lateral uterine walls and involving the region of the parametria .

ELIGIBILITY:
Inclusion Criteria:

All patients diagnosed with placenta previa previa or low lying placenta during pregnancy at any gestational age will be included and followed up until termination of pregnancy. The diagnosis of placenta previa was based on the presence of placental tissue overing the internal cervical os and Low-lying placenta was diagnosed when the placenta was within 2 cm from the internal cervical os but did not cover it

Exclusion Criteria:

* Impaired liver or renal functions.
* Coagulation disorders.
* Associated uterine pathology needing hysterectomy.
* Patient's refusal to participate in clinical research.
* Multiple pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: All females in age range between 18 years old and 45 years old who are diagnosed as placenta accreta spectrum disorder in antenatal care at Assiut University, Women Health Hospital at time between May 2021 and May 2023 will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate the association of ultrasonographic parameters with the intraoperative FIGO clinical grading for diagnosis of placenta accreta spectrum disorder and histopathological diagnosis of placenta accreta in hysterectomy specimens | Bseline
  Grade 1 : Complete placental separation at third stage, Grade 2 : removal of placenta required and parts of placenta thought to be abnormally adherent, Grade 3 : Manual removal of placenta required and the whole placental bed thought to be abnormally adherent, Grade 4 : Placental tissue seen to have invaded through the serosa of the uterus but a clear surgical plane can be identified between the bladder and uterus, Grade 5 : Placental tissue seen to have invaded through the serosa of the uterus and a clear surgical plane cannot be identified between the bladder and uterus, Grade 6 : Placental tissue seen to have invaded through the serosa of the uterus and infiltrating the parametrium or any organ other than the urinary bladder

SECONDARY OUTCOMES:
Association of each ultrasonographic parameter of placental invasion with maternal and fetal complications | Baseline
  1. Maternal complications both intra and post-operatively including cesarean hysterectomy, ICU admission, bladder injury, bowel injury and death.
  2. Fetal and neonatal complications including Apgar score less than 7 at 5 min, RDS, NICU, preterm and neonatal death.
  3. Development of ultrasound scoring system for prediction of placenta accreta.

IPD SHARING:
Plan to Share IPD: Undecided